CLINICAL TRIAL: NCT05859971
Title: Use of ICG-fluorescent Imaging for Sentinel Lymph Node Mapping in Patients With Breast Cancer
Brief Title: ICG and SLN Mapping
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: OnLume Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-0030; 5R44CA206754 (NIH); UW22145 (Other: UW Madison); SMPH/SURGERY/SURG ONC (Other: UW Madison); Protocol Version 11/29/2022 (Other: UW Madison)
Record Dates: First submitted 2023-04-06; First posted 2023-05-16 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; sentinel lymph node; ICG fluorescence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Sentinel Lymph Node (SLN) mapping (Experimental): SLN mapping and biopsy will be performed using technetium-99m sulfur colloid and isosulfan blue dye, as well as ICG-fluorescent imaging.
  Interventions: Drug: SLN mapping using technetium-99m +/- isosulfan blue dye; Device: SLN mapping with ICG fluorescence using the Asimov Platform

INTERVENTIONS:
Drug: SLN mapping using technetium-99m +/- isosulfan blue dye — The isosulfan blue dye injection will be performed by the participating surgeon in the operating room; as per standard of care, injection will be subareolar. Incisions will be planned based on the technetium-99m activity or at the lateral aspect of the pectoralis muscle, per usual care.
Device: SLN mapping with ICG fluorescence using the Asimov Platform — 2 ml (5 mg) of ICG solution will be injected intradermally in 1-4 injection sites in the lateral areolar region. After injection, gentle manual massage will be performed for 5 minutes. ICG imaging will be obtained prior to incision. After incision is made (following standard of care procedures), the axilla will be visualized using the Asimov Platform to assess for ICG-fluorescence in sentinel lymph nodes.

SUMMARY:
The purpose of this research study is to assess the feasibility of using a different dye and imaging device, indocyanine green (ICG)-fluorescent imaging through the Asimov Imaging Platform, to perform sentinel lymph node biopsy.

Participants in this research study will be undergoing a sentinel lymph node biopsy as part of surgical treatment for breast cancer. Active participation will last through the post-operative visit.

DETAILED DESCRIPTION:
In this study, the sentinel lymph node biopsy will be performed with radioactive tracer (technetium-99 sulfur colloid) and blue dye, which is standard of care. Decisions will be made during surgery about which lymph nodes to remove using information from the radioactive tracer and blue dye alone.

For this research, ICG fluorescence dye during participant's surgery will also be used. After anesthesia has started, the ICG fluorescence dye will be injected in the breast along at the edge of the areola in the same location as the radioactive tracer and blue dye injections. The breast and axilla will then be imaged with the Asimov Imaging Platform to look for the sentinel lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosis of clinical T1 or T2 breast cancer clinically node negative breast cancer requiring surgical lymph node evaluation
* Surgery at University of Wisconsin Hospital and Clinic

Exclusion Criteria:

* Pregnant: It is not known whether indocyanine green can cause fetal harm when administered to a pregnant woman or can affect reproduction capacity. Women of child-bearing age will undergo a urine pregnancy test on the day of surgery, which is standard of care prior to anesthesia.
* Breastfeeding: It is not known whether this drug is excreted in human milk. Because many drugs are excreted in human milk, caution should be exercised when indocyanine green is administered to a nursing woman. Study team will exclude women who are breastfeeding.
* Unable to provide informed consent
* Allergy to indocyanine green
* History of ipsilateral breast or axillary surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Neuman, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in April and May of 2023.
Period: Overall Study
Arm/Group | Sentinel Lymph Node (SLN) Mapping
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sentinel Lymph Node (SLN) Mapping
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 60.8 [45 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Concordance Between Detection of Sentinel Lymph Nodes by ICG Versus Technetium-99, at the Lymph Node Level
Description: The study team will describe concordance rates between technetium-99 and ICG-fluorescence for each sentinel lymph node removed.
Time Frame: Day of operation
Measure: Number; unit: percent concordance
Arm/Group | Sentinel Lymph Node (SLN) Mapping
Number analyzed (Participants) | 10
percent concordance | 100

2. Primary Outcome: Concordance Between Detection of Sentinel Lymph Nodes by ICG Versus Technetium-99, at the Patient Level
Description: The study team will assess concordance rates at the patient level rates between technetium-99 and ICG-fluorescence.
Time Frame: Day of operation
Measure: Number; unit: percent concordance
Arm/Group | Sentinel Lymph Node (SLN) Mapping
Number analyzed (Participants) | 10
percent concordance | 100

3. Secondary Outcome: Accuracy of the ICG Mapping
Description: Using the technetium-99as the gold standard, the study team will describe the number of lymph nodes that would have been missed (i.e. technetium-99 + but ICG- in removed SLN) or would have been excised unnecessarily (i.e. residual ICG-fluorescence in axilla but no residual technetium-99) if ICG-fluorescent imaging had guided the SLN.
Time Frame: Day of operation
Population: unable to assess, see post-hoc measures for data available and limitations and caveats for relevant detail
Arm/Group | Sentinel Lymph Node (SLN) Mapping
Number analyzed (Participants) | 0

4. Post Hoc Outcome: Number of Participants With Residual Radioactivity
Time Frame: Day of operation
Measure: Count of Participants; unit: Participants
Arm/Group | Sentinel Lymph Node (SLN) Mapping
Number analyzed (Participants) | 10
Participants | 10

5. Post Hoc Outcome: Number of Participants With Visible Fluorescence in the Axilla
Time Frame: day of operation
Measure: Count of Participants; unit: Participants
Arm/Group | Sentinel Lymph Node (SLN) Mapping
Number analyzed (Participants) | 10
Participants | 8

ADVERSE EVENTS:
Time Frame: Through post-operative visit, up to 3 weeks
Arm/Group | Sentinel Lymph Node (SLN) Mapping
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Difficult to differentiate general staining of the tissue from the ICG versus true residual fluorescence in a lymph node.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT05859971/Prot_SAP_000.pdf